CLINICAL TRIAL: NCT01535846
Title: Awakening to the Taste of Food: What Are the Effects on Cognitions and Behaviors About Food and Eating Among Restrained Women?
Brief Title: Awakening to the Taste of Food Among Restrained Women
Acronym: Flaveur
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Foundation for Dietetic Research (CFDR) (Other)
Responsible Party: Principal Investigator, Véronique Provencher, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: INAF 2010-215
Record Dates: First submitted 2012-02-13; First posted 2012-02-20 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Other Eating Disorders
Keywords: taste; mindful eating; intuitive eating; attitude; behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conscious food tasting intervention (Experimental): Instead of focusing on dieting rules to restrict food intake, paying attention to sensory stimulation allow the recognition of internal cues of hunger and satiety which can be helpful to facilitate a more internalized regulation of food intake among restrained eaters. In the experimental group, the conscious food tasting intervention will be conducted by a registered dietitian into small groups of ten to twelve women during six weekly 2-hour workshops. Workshops will be taking place in a well-ventilated room to insure that there are no extraneous odours or noises that may hamper the activities involving senses.
  Interventions: Behavioral: Conscious food tasting intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Conscious food tasting intervention — Six weekly 2-hour workshops
  Arms: Conscious food tasting intervention

SUMMARY:
Energy-restricted diets often require dieting rules, which forced the dieter to eat according to cognitive norms, which increase his vulnerability to external food cues. Allowing the recognition of internal hunger and satiety cues by using conscious food tasting could be helpful among restrained eaters to facilitate an internalized regulation of food intake.

The objectives of the proposed study are to investigate among restrained women whether conscious food tasting can influence 1) attitudes and behaviors associated with food and eating; 2) reliance on hunger and satiety signals; and 3) development of taste and olfactory memory.

Females (n=50) will be randomly assigned to: 1) experimental group (conscious food tasting intervention) (n=24), or 2) control group (n=26). The conscious food tasting intervention will be conducted by a registered dietitian into groups of ten to twelve women during six weekly 2-hour workshops. Women in the control group will not receive any intervention. Measurements will be taken at baseline, at the end of the intervention period, and at 12-week post-intervention. Restraint Scale, Three-Factor Eating Questionnaire, Mindful Eating Questionnaire, Intuitive Eating Scale, Body-Esteem Scale and Rosenberg Self-Esteem Scale will measure attitudes and behaviors associated with food and eating as well as some aspects related to psychological functioning. The Intuitive Eating Scale and a snack-meal taste rating task (visual analogue scales) will assess internal hunger/satiety cues. Vocabulary used to describe the foods will be recorded from the snack-meal taste rating task and use to assess taste and olfactory memory. Sensory capabilities will be assessed by odour detection and identification test, and a taste detection test.

The proposed study will provide a better understanding of the effects of conscious food tasting on eating attitudes and behaviors, which is relevant to dietetic practice as it could help to promote sustainable healthy eating habits.

DETAILED DESCRIPTION:
In the experimental group (n=24), the conscious food tasting intervention will be conducted by a registered dietitian into small groups of ten to twelve women during six weekly 2-hour workshops. Workshops will be taking place in a well-ventilated room to insure that there are no extraneous odours or noises that may hamper the activities involving senses. To enhance feeling of belonging to the group as well as the confidence within each participant, time will be allowed for participants' introduction at the beginning of the first workshop. Specific themes will be addressed during each of the six workshops. During the first and second workshops, theoretical notions about weight management and energy-restricted diets, restrained eating versus intuitive and mindful eating, appetite sensations, sensory-specific satiety and weight-related issues will be presented by the registered dietitian. The presentation will be interactive, so that discussion and questions will be foster throughout the workshops. From the third workshop, basic knowledge and activities related to sensory food perceptions will be introduced. Prior to food tasting activities, participants will be advised to avoid drinking coffee or eating chocolate and any other foods with a strong or persistent taste, and to avoid wearing perfumes, scented lotions and creams as all these conditions could affect sensory perceptions. During the third workshop, theoretical notions about taste qualities (sweet, salt, sour, bitter) will be firstly addressed. A taste activity will then be done using aqueous solutions containing different concentrations of a taste compound. The objective of this activity will be to let participants experience their own taste sensitivity level so that they can identify at which concentration level they can detect different tastes. During the fourth and fifth workshop, theoretical and practical notions about food tasting techniques will be addressed. The various roles played by other senses (i.e., sight, hearing, touch, smell) during food tasting will also be experienced by the participants using practical activities. For that purpose, various foods will be used such as herbs and spices, cheeses, fruits, chocolate and chips. In addition, one of the most difficult aspects of tasting evaluation is to find the right words that well-described food perception. Each participant will thus be guided by the registered dietitian and discuss about some of the terminology of tasting in order to find out appropriate terms they could be used to describe the tasted foods. A list of these descriptive words will then be created, so that they can have their own list of reference. At the end of each food tasting activities, a discussion will be led by the registered dietitian about appetite sensations, emotions and recollection of memories associated with the tasted foods. As enjoying eating involve more than sensory stimulation from the foods, the last workshop will discuss the cognitive, social and emotional aspects related to tasting and pleasure while eating (e.g. dichotomized thinking about healthy eating, eating with family and friends, and affective processes in eating behaviors) in order to integrate these eating-related aspect to a peaceful relationship with foods.

In the waiting-list control group (n=26), women will be instructed to follow their usual lifestyle habits for the duration of the study. Over the study period, these women will not receive any form of contact from the research team, with the exception of post treatment testing sessions (T=2 and T=3), as performed in the experimental group. To control for potential confounding effects of other treatments, the investigators will ask to women from the waiting-list control group to report all consultations with health professionals and/or any forms of intervention that they received during the course of the study. After the final testing session at 12-week post-intervention (T=3), women from the control group will be invited to participate in the conscious food tasting intervention on a voluntary basis.

ELIGIBILITY:
Inclusion Criteria:

* females aged 25 to 60 year-old
* stable weight (± 2.5 kg) for at least 2 months
* restrained eaters (scores of 15 or higher at the Restraint Scale)

Exclusion Criteria:

* food allergies
* taking medication (e.g., corticosteroids, tricyclic antidepressants, atypical antipsychotics)
* chronic health problems (e.g., eating disorders, type 1 and type 2 diabetes, hyperthyroidism)
* pregnant or lactating
* smoker

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Attitudes and behaviors associated with food and eating | Up to 3 months
  To evaluate the effects of conscious food tasting on attitudes and behaviors associated with food and eating. This measure is made through a questionnaire.

SECONDARY OUTCOMES:
Physical signals for hunger and satiety | Up to 3 months
  To assess whether conscious food tasting affect reliance on physical signals for hunger and satiety (rather than external cues). This measure is made through a questionnaire.
Development of taste and olfactory memory | Up to 3 months
  To evaluate the effects of conscious food tasting on the development of taste and olfactory memory. This measure is made through a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Provencher, Ph.D., Principal Investigator — Laval University
Locations (1):
- Institute of Nutraceuticals and Functionnal Foods (INAF), Québec, Quebec, Canada